CLINICAL TRIAL: NCT01313585
Title: Retrospective, Real-life Observational Evaluation of the Effectiveness of Mixed Maintenance and Reliever Inhaler Types in Patients in the Management of Asthma in a Representative UK Primary Care Population
Brief Title: Device Mixing in Asthma, a General Practice Research Database Study
Acronym: EBsalbutamol
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Professor David Price, Research in Real Life
Other Study IDs: 003/10
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Asthma
Keywords: Primary care; asthma management; inhaler device; maintenance therapy; reliever therapy; Easibreathe salbutamol
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- IPDA salbutamol MDI: receive a recorded increase in ICS therapy as BDP Easibreathe at the index date and also receive salbutamol MDI
  Interventions: Drug: Increase of beclometasone via the Easibreathe device plus salbutamol via an MDI
- IPDA salbutamol EB: receive a recorded increase in ICS therapy as BDP Easibreathe at the index date and also receive salbutamol Easibreathe
  Interventions: Drug: Increase of beclometasone via the Easibreathe device plus salbutamol via the Easibreathe device
- IPDI salbutamol EB: initiate ICS therapy as BDP Easibreathe at the index date and also receive salbutamol Easibreathe
  Interventions: Drug: Initiation of beclometasone via the Easibreathe device plus salbutamol via the Easibreathe device
- IPDI salbutamol MDI: initiate ICS therapy as BDP Easibreathe at the index date and also receive salbutamol MDI
  Interventions: Drug: Initiation of beclometasone via the Easibreathe device plus salbutamol via and MDI device

INTERVENTIONS:
Drug: Initiation of beclometasone via the Easibreathe device plus salbutamol via the Easibreathe device
  Groups: IPDI salbutamol EB
Drug: Initiation of beclometasone via the Easibreathe device plus salbutamol via and MDI device
  Groups: IPDI salbutamol MDI
Drug: Increase of beclometasone via the Easibreathe device plus salbutamol via the Easibreathe device
  Groups: IPDA salbutamol EB
Drug: Increase of beclometasone via the Easibreathe device plus salbutamol via an MDI
  Groups: IPDA salbutamol MDI

SUMMARY:
This study will compare the absolute and relative effectiveness of asthma management in patients on inhaled corticosteroid (ICS) maintenance therapy as Easi-breathe® (EB) - beclometasone dipropionate (BDP) breath-actuated inhaler (BAI) - and as-needed (prn) reliever medication (short-acting beta2-agonist [SABA] therapy) via either a BAI (i.e. Easi-breathe® [EB] salbutamol) or via a pressurised metered dose inhaler (MDI) (e.g. MDI salbutamol).

DETAILED DESCRIPTION:
Current asthma guidelines in the UK are underpinned by evidence derived from randomised controlled trials (RCTs). Although RCT data are considered the gold standard, patients recruited to asthma RCTs are estimated to represent less than 10% of the UK's asthma population. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is, therefore, a need for more representative RCTs and real-life observational studies to inform existing guidelines and help optimise asthma outcomes.

Inhalation therapy is the cornerstone of asthma treatment, used for the delivery of 'reliever' bronchodilator therapy (e.g. salbutamol) as well as anti-inflammatory corticosteroid 'maintenance' or 'controller' therapy. Currently available inhaler devices include MDIs, breath-actuated MDIs (BAIs), and dry powder inhalers (DPIs). Both BAIs and DPIs are actuated by the patient's inhalation manoeuvre, while MDIs are actuated by the patient's pressing of a button, which must thus be coordinated with inhalation. The clinical effectiveness of inhalation therapy derives from delivery of drug to the target sites in the lungs, and evidence is mounting that suboptimal use of inhaler devices is a common problem contributing to compromised asthma control for many patients. Indeed, decreased asthma control has been linked to the number of mistakes when using MDIs for delivering inhaled corticosteroids (ICS).

There is also evidence that the ability of patients to use the different inhaler device types is variable. Nonetheless, recent reviews of RCTs, while recognising the importance of inhaler technique, have concluded that inhaler devices do not differ significantly in efficacy and that the cheapest inhaler device should be used. However, as results are based on RCTs they should be applied with care in light of the aforementioned issues around external validity of RCTs and the ability to extrapolate their findings across a broad patient population. Moreover, patients enrolled in RCTs typically receive extensive training and must demonstrate and maintain proper inhaler technique, seldom accomplished in a real-world setting.

The aim of this study is to compare the absolute and relative effectiveness of ICS (maintenance) plus SABA (reliever) therapy delivered via same-type devices (namely BDP via EB plus salbutamol via EB [BAI]) and that delivered via different device types (i.e. BDP via EB [BAI] plus SABA via MDI) in a real-life, representative, UK primary care asthma population.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 4-80 years:

  * Paediatric cohort (aged 4-11 years), and
  * Adult cohort (aged 12-80 years )
* Evidence of asthma:

  * a diagnostic code for asthma, and / or
  * ≥2 prescriptions for asthma at different points in time during the prior year and/ or
  * ≥2 prescriptions for asthma therapies during the outcome year, including ≥1 ICS prescription (in addition to that received at IPD) - IPDI cohort only
* Be on current asthma therapy (for the IPDA cohort only):

  * ≥1 ICS prescription in the prior year, and
  * ≥1 other asthma prescription during the baseline year.
* Have at least one year of up-to-standard (UTS) baseline data (prior to the IPD) and at least one year of UTS outcome data (following the IPD).

Exclusion Criteria:

* had a COPD read code at any time; and/or
* received a combination inhaler in addition to a separate ICS inhaler in the baseline year; and/or
* received a long-acting beta2-agonsist (LABA) in addition to a separate ICS inhaler in the baseline year
* received ICS therapy during baseline year via DPI (in IPDA cohort only).

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthma patients on SABA therapy (any available) monotherapy who, at the index date, either:
  (i) IPDI: initiate ICS therapy as BDP EB at the index date and also receive reliever therapy as either*:
  * Salbutamol EB, or
  * Salbutamol MDI, OR, who (ii) IPDA: receive a recorded increase in ICS therapy as BDP EB at the index date and also receive reliever therapy as either*:
  * Salbutamol EB, or
  * Salbutamol MDI.
Sampling Method: Non-Probability Sample
Enrollment: 815377 (Actual)
Dates: Start 1991-01; Primary Completion 2007-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Proxy asthma control | One-year outcome period
  Control defined as:
  * No recorded hospital attendance for asthma, including admission, Accident & Emergency (A&E) attendance, out-of-hours attendance, or Out-Patient Department (OPD) attendance, AND
  * No prescriptions for oral steroids, AND
  * No GP consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics.
Total number of asthma exacerbations and exacerbation rate ratio | One-year outcome period
  Where exacerbation is defined as an occurrence of:
  * Unscheduled hospital admissions / A&E attendance for asthma, OR
  * Use of oral steroids

SECONDARY OUTCOMES:
Treatment success 1 | One-year outcome period
  Success: defined as:
  (i) Exacerbation:
  1. Unscheduled hospital admissions / A&E attendance for asthma, OR
  2. Acute use of oral steroids
  AND
  (ii) No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics
  AND
  (iii) No change in therapeutic regimen:
  1. Increased dose of ICS, and/or
  2. Change in ICS/LABA, and/or
  3. Change in delivery device, and/or
  4. Use of additional therapy as defined by: theophylline, leukotreine receptor antagonists (LTRAs).
Treatment success 2 (independent of possible cost savings) | One-year outcome period
  Success: defined as:
  (i) Exacerbation:
  1. Unscheduled hospital admissions / A&E attendance for asthma, OR
  2. Acute use of oral steroids
  AND
  (ii) No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics
  AND
  (iii) No change in therapeutic regimen:
  1. Increased dose of ICS, and/or
  2. Use of additional therapy as defined by: theophylline, leukotreine receptor antagonists (LTRAs).
Respiratory-related hospitalisations and referrals. | One-year outcome period
  Mean number of respiratory-related hospitalisations and referrals per patient recorded during the one-year outcome period

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof. MD, Principal Investigator — Company Director; Alison Chisholm, MSc, Study Director — Research Project Director
Locations (1):
- General Practice Research Database, London, London, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Cohort Health Study Team. Spirometric criteria for asthma: adding further evidence to the debate. J Allergy Clin Immunol. 2005 Nov;116(5):976-82. doi: 10.1016/j.jaci.2005.08.034. PMID 16275363
- [Background] Crompton GK, Barnes PJ, Broeders M, Corrigan C, Corbetta L, Dekhuijzen R, Dubus JC, Magnan A, Massone F, Sanchis J, Viejo JL, Voshaar T; Aerosol Drug Management Improvement Team. The need to improve inhalation technique in Europe: a report from the Aerosol Drug Management Improvement Team. Respir Med. 2006 Sep;100(9):1479-94. doi: 10.1016/j.rmed.2006.01.008. Epub 2006 Feb 21. PMID 16495040
- [Background] Chrystyn H, Price D. Not all asthma inhalers are the same: factors to consider when prescribing an inhaler. Prim Care Respir J. 2009 Dec;18(4):243-9. doi: 10.4104/pcrj.2009.00029. PMID 19513494
- [Background] Giraud V, Roche N. Misuse of corticosteroid metered-dose inhaler is associated with decreased asthma stability. Eur Respir J. 2002 Feb;19(2):246-51. doi: 10.1183/09031936.02.00218402. PMID 11866004
- [Background] Lenney J, Innes JA, Crompton GK. Inappropriate inhaler use: assessment of use and patient preference of seven inhalation devices. EDICI. Respir Med. 2000 May;94(5):496-500. doi: 10.1053/rmed.1999.0767. PMID 10868714
- [Background] Molimard M, Raherison C, Lignot S, Depont F, Abouelfath A, Moore N. Assessment of handling of inhaler devices in real life: an observational study in 3811 patients in primary care. J Aerosol Med. 2003 Fall;16(3):249-54. doi: 10.1089/089426803769017613. PMID 14572322
- [Background] Brocklebank D, Ram F, Wright J, Barry P, Cates C, Davies L, Douglas G, Muers M, Smith D, White J. Comparison of the effectiveness of inhaler devices in asthma and chronic obstructive airways disease: a systematic review of the literature. Health Technol Assess. 2001;5(26):1-149. doi: 10.3310/hta5260. PMID 11701099
- [Background] Brocklebank D, Wright J, Cates C. Systematic review of clinical effectiveness of pressurised metered dose inhalers versus other hand held inhaler devices for delivering corticosteroids in asthma. BMJ. 2001 Oct 20;323(7318):896-900. doi: 10.1136/bmj.323.7318.896. PMID 11668133
- [Background] Dolovich MB, Ahrens RC, Hess DR, Anderson P, Dhand R, Rau JL, Smaldone GC, Guyatt G; American College of Chest Physicians; American College of Asthma, Allergy, and Immunology. Device selection and outcomes of aerosol therapy: Evidence-based guidelines: American College of Chest Physicians/American College of Asthma, Allergy, and Immunology. Chest. 2005 Jan;127(1):335-71. doi: 10.1378/chest.127.1.335. PMID 15654001
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org